CLINICAL TRIAL: NCT03054467
Title: Effect of Amlodipine Versus Amlodipine Combined With Atorvastatin on the Symptoms, Function, and Quality of Life in Patients With Coronary Vasospastic Angina
Brief Title: Effect of Amlodipine Versus Amlodipine Combined With Atorvastatin on the Coronary Vasospastic Angina
Acronym: SCARLET
Status: Unknown | Phase: Phase 4 | Type: Interventional
Last Known Status: Not yet recruiting
Sponsor: Kosin University Gospel Hospital (Other)
Responsible Party: Principal Investigator, Kyoung Im Cho, Associate Professor, Kosin University Gospel Hospital
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: SCARLET
Record Dates: First submitted 2017-02-12; First posted 2017-02-15 (Actual); Last update posted 2018-08-10 (Actual); Status verified 2018-08

CONDITIONS: Quality of Life
MeSH Terms: interventions — amlodipine, atorvastatin drug combination; Amlodipine

STUDY DESIGN:
Who Masked: Participant, Investigator
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- CADUET 10mg-20mg (Active Comparator): Patients are assigned to receive either amlodipine therapy (NORVASC 10 mg/day) for 6 months.
  Interventions: Drug: Caduet 10Mg-20Mg Tablet
- NORVASC (Active Comparator): Patients are assigned to receive amlodipine/atorvastatin combination (CADUET 10/20mg) for 6 months
  Interventions: Drug: NorvasC® 10 mg Tablets

INTERVENTIONS:
Drug: Caduet 10Mg-20Mg Tablet — Patients are randomly assigned to receive either amlodipine therapy (NORVASC 10 mg/day) or amlodipine/atorvastatin combination (CADUET 10/20mg) for 6 months. The starting dose of the drung is either 5mg amlodipine or 5/20mg CADUET. After 4 weeks, if the 5mg amlodipine is well tolerated, the dose is titrated to 10mg and 10/20mg CADUET
  Arms: CADUET 10mg-20mg
Drug: NorvasC® 10 mg Tablets — Patients are randomly assigned to receive either amlodipine therapy (NORVASC 10 mg/day) or amlodipine/atorvastatin combination (CADUET 10/20mg) for 6 months. The starting dose of the drung is either 5mg amlodipine or 5/20mg CADUET. After 4 weeks, if the 5mg amlodipine is well tolerated, the dose is titrated to 10mg and 10/20mg CADUET
  Arms: NORVASC

SUMMARY:
The aim of the present study is to compare the effects of CCB and CCB+ high dose of statin therapy on the symptoms, function, and quality of life assessed by validated angina-specific questionnaire (Short-form Seattle Angina Questionnaire (SAQ-7)), endothelial function as measured by FMD of the brachial artery, endothelial progenitor cells (EPC) and coronary flow reserve (CFR) in patients with VSA.

DETAILED DESCRIPTION:
STUDY DESIGN Study protocol Study Start (expected FSFV (First subject first visit )) at August 1 2016 Study Stop (expected LSLV (Last subject last visit)) at February 29 2019 150 Patients with confirmed VSA who had over 3 episodes of angina per week during a over 2 week qualification period are randomly assigned to receive either amlodipine therapy (NORVASC 10 mg/day) or amlodipine/atorvastatin combination (CADUET 10/20mg) for 6 months. The starting dose of the drung is either 5mg amlodipine or 5/20mg CADUET. After 4 weeks, if the 5mg amlodipine is well tolerated, the dose is titrated to 10mg and 10/20mg CADUET. All other antianginal medications are proscribed during the study period except long-acting nitrates and sublingual nitroglycerin as required. Long-acting nitrates are permitted during the study period if they had been taken at a constant dosage for over 2 weeks before study entry. Participants are allowed to take sublingual NTG as needed for episodes of chest pain.

Study design. Patients with VSA who had over 1 angina episodes/week confirmed by ergonovine provocation test Acquisition of written consent Randomization to NORVASC 10 mg/day or CADUET 10/20 mg Baseline SAQ, angina diary, FMD, EPC, CFR assessments are performed. Medication start with either 5mg NORVASC or 5/20mg CADUET. After 4 weeks, if the 5mg amlodipine is well tolerated, titrate to 10mg and 10/20mg CADUET. Routine visit with the scheduled reservation (2 or 3 months interval) After 6-months treatment, follow-up SAQ, angina diary, FMD, EPC, CFR assessments are performed (mandatory).

After 12-months treatment, follow-up SAQ, angina diary, FMD, EPC, CFR assessments are performed (optional).

Efficacy assessments. The primary efficacy variable is the change of summary score of SAQ-7 between NORVASC 10mg/day and CADUET 10/20mg, and the weekly average frequency of self-reported angina episodes during the 6-months treatment phase. Difference of Summary score of SAQ 7 is calculated between the baseline (at the enrollment before randomization) and the after 6-months treatment. The study staff at each clinical site will review the angina and nitroglycerin use diaries with the patient at each study visit.

Assessment of patient responses by short form SAQ at baseline and after 6 months treatment.

The Seattle Angina Questionnaire (SAQ) is a validated disease-specific instrument for assessing the health status of patients with coronary artery disease. Although the SAQ has been frequently used in clinical trials and registries, its use in routine clinical care has been limited by its length (19 questions) and the absence of a single summary score that facilitates an overall assessment of patients' health status.

Recently, 7-item from the Physical Limitation, Angina Frequency, and Quality of Life domains for the shortened version of the SAQ (SAQ 7), as well as an overall summary score was developed and validated in patients with stable coronary artery disease, undergoing percutaneous coronary intervention, and presenting with acute myocardial infarction.

ELIGIBILITY:
* The investigators include patients who are newly diagnosed with VSA within 3 months of the screening and patients without CCB during the 1month of screening.
* VSA patients who had over 3 episodes of angina per week during a over 2-week qualification period will be included.
* In addition to the angina symptoms, the following two criteria for diagnosing VSA needed to be satisfied:

  * (1) spontaneous or ergonovine induced coronary artery spasm (producing over 90% narrowing of coronary lumen diameter during angiography) associated with chest pain and ischemic ST segment changes (transient ST elevation or depression over 0.1 mV, recorded from at least two contiguous leads on the 12-lead ECG);
  * (2) normal or insignificant (diameter stenosis under 50%) coronary artery disease after intracoronary nitroglycerine injection.
* The investigators exclude patients who have fixed stenosis corresponding to ≥50% of the lumen diameter in the coronary artery and those who have a history of allergic reaction to amlodipine or atorvastatin.
* Other exclusion criteria are:

  * (1) myocardial infarction within 3 months of screening;
  * (2) history of life threatening events associated with previous episodes of coronary artery spasm, such as ventricular tachycardia, ventricular fibrillation, or syncopal episodes;
  * (3) decompensated congestive heart failure;
  * (4) significant valvular heart disease;
  * (5) systolic blood pressure under 90 mm Hg;
  * (6) baseline heart rate over 100 beats/min;
  * (7) ECG abnormalities precluding interpretation of the ST changes;
  * (8) coronary artery bypass surgery or percutaneous coronary intervention within 3 months of screening;
  * (9) women of childbearing potential who refused to use contraception;
  * (10) active hepatic or renal disease;
  * (11) other major concomitant disease.

Ages: 18 Years to 70 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 150 (Estimated)
Dates: Start 2018-12-01 (Estimated); Primary Completion 2019-04-28 (Estimated); Study Completion 2019-04-28 (Estimated)

PRIMARY OUTCOMES:
Overall summary score assessed by short form SAQ | 6 months

SECONDARY OUTCOMES:
FMD of the brachial artery | 6 months
The change of Coronary flow reserve (CFR) assessed in the dLAD using TTE | 6 months
Angina frequency from the patient's diary | 6 months
Measurements of circulating endothelial progenitor cells (EPCs) | 6 months

IPD SHARING:
Plan to Share IPD: No